CLINICAL TRIAL: NCT04623801
Title: Pilot Study to Evaluate the Safety and Efficacy of Percutaneous Laser Ablation of Thyroid Papillary Microcarcinoma
Brief Title: Laser Ablation of Papillary Thyroid Microcarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-438
Record Dates: First submitted 2020-11-06; First posted 2020-11-10 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Papillary Thyroid Microcarcinoma; Thyroid; Thyroid Cancer
Keywords: PTMC; Papillary Thyroid Microcarcinoma; Thyroid Cancer; Percutaneous Laser Ablation; PLA; 19-438; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma; Thyroid Diseases; Thyroid Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with papillary microcarcinoma (PTMC) (Experimental): Participants with papillary microcarcinoma (PTMC) who have elected to proceed with thyroidectomy rather than an observational management approach will be considered as potential candidates for this trial.
  Interventions: Procedure: Percutaneous Laser Ablation (PLA)

INTERVENTIONS:
Procedure: Percutaneous Laser Ablation (PLA) — Percutaneous Laser Ablation / PLA will be carried out in a single session by advancing one 21-gauge spinal needle into the target lesions under real time US guidance.

SUMMARY:
The purpose of this study is to explore whether percutaneous laser ablation (PLA) is a safe and effective alternative to removing papillary thyroid microcarcinoma (PTMC) with surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Papillary thyroid cancer documented by

  * (a) Bethesda VI cytology,
  * (b) Bethesda III, IV, V, or VI cytology AND BRAF V600E mutation, or
  * (c) Bethesda V cytology AND high risk ultrasonographic features documented by either the ATA high suspicion or TIRADS 5 nodule characteristics

To ensure the majority of cases will be eligible based on criteria (a) or (b), we will enroll ≤ 2 patients based on criteria (c).

* Maximum diameter ≤ 13 mm
* Declined active surveillance
* The thyroid lesion must be primarily solid with ≤ 25% cystic compent
* No US evidence of extrathyroidal extension through the thyroid capsule
* No imaging evidence of lymph node metastasis
* Preserved contralateral vocal cord function prior to PLA

Exclusion Criteria:

* Thyroid cancer that is non papillary thyroid cancer (PTC)
* Thyroid lesion with > 25% cystic component
* Lesion with US evidence of extrathyroidal extension through the thyroid capsule
* Clinical or ultrasonographic evidence of lymph node metastasis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete thermal ablation | 6 months
  Complete thermal ablation of the targeted PTMC (T1aN0M0) as determined by histological examination of thyroid tissue obtained by either thyroid lobectomy or total thyroidectomy 6 months after PLA.

CONTACTS AND LOCATIONS:
Overall Officials: R. Michael Tuttle, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org